CLINICAL TRIAL: NCT04305249
Title: A Phase I, Open-Label, Multi-Center Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG-017 Monotherapy or Combination Therapy With Nivolumab in Patients With Advanced Solid Tumors and Hematological Malignancies
Brief Title: Safety and Preliminary Efficacy of ATG-017 Monotherapy or Combination Therapy With Nivolumab in Advanced Solid Tumors and Hematological Malignancies
Acronym: ERASER
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on the internal need to re-prioritization the whole pipeline and phase 1 portfolio.
Sponsor: Antengene Therapeutics Limited (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-017-001
Record Dates: First submitted 2020-03-05; First posted 2020-03-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module A (ATG-017 Monotherapy) (Experimental): Dosing will begin at 5 mg QD ATG-017 as starting dose. A treatment cycle will be 21 days for continuous dosing and 28 days for 7 days on/7 days off intermittent dosing of ATG-017 treatment.
  Interventions: Drug: ATG-017
- Module B (ATG-017+Nivolumab Combination Therapy in Solid Tumors) (Experimental): With the combination with nivolumab, a cycle of study treatment will be defined as 28 days. ATG-017 is planned initially to be continuously given 28 days in each cycle. ATG-017 dosing schedule in combination therapy will follow a similar dose escalation principle as with monotherapy but starting at 5 mg BID. Nivolumab will be given at fixed dosing, 480 mg Q4W, on D1 of each cycle.
  Interventions: Drug: ATG-017+Nivolumab

INTERVENTIONS:
Drug: ATG-017 — Dosing will begin at 5 mg QD ATG-017 as starting dose. A treatment cycle will be 21 days for continuous dosing and 28 days for 7 days on/7 days off intermittent dosing of ATG-017 treatment.
  Other Names: AZD0364 hemi-adipic acid
  Arms: Module A (ATG-017 Monotherapy)
Drug: ATG-017+Nivolumab — With the combination with nivolumab, a cycle of study treatment will be defined as 28 days. ATG-017 is planned initially to be continuously given 28 days in each cycle. ATG-017 dosing schedule in combination therapy will follow a similar dose escalation principle as with monotherapy but starting at 5 mg BID. Nivolumab will be specified dose on specified days.
  Other Names: AZD0364 hemi-adipic acid+Opdivo
  Arms: Module B (ATG-017+Nivolumab Combination Therapy in Solid Tumors)

SUMMARY:
This is a Phase I, multi-center, open-label study of ATG-017 administered orally, alone or in combination with nivolumab in patients with advanced solid tumors and hematological malignancies. The study is composed of two modules: ATG-017 monotherapy (Module A) and ATG-017 in combination with nivolumab (Module B). Both Modules A and B will include Dose Escalation Phase and Dose Expansion Phase.

DETAILED DESCRIPTION:
The dose escalation of ATG 017 will be conducted with intensive safety monitoring to ensure the safety of the patients with solid tumors (Module A and Module B) and hematological malignancies (Module A) harbouring activating alterations in the RAS-MAPK pathway, and will include the continuous and intermittent dosing schedules.

The Dose Expansion Phase will start based on dose level and schedule (continuous or intermittent)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
2. Aged at least 18 years.
3. Module A: Patient must have a documented activating alteration of the RAS-MAPK pathway.
4. Module B: Dose Escalation Phase: Patient must have a documented activating alteration of the RAS-MAPK pathway; Dose Expansion Phase: Expansion cohorts will be further defined based on information from the Dose Escalation.
5. Histological or cytological confirmation of a solid tumour.
6. Patient with solid tumors must have at least 1 lesion, not previously irradiated.
7. Estimated life expectancy of minimum of 12 weeks.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
9. Ability to swallow and retain oral medication.

Exclusion Criteria:

1. Central nervous system metastatic disease, leptomeningeal disease, or metastatic cord compression.
2. Prior ATG-017 administration in the present study.
3. Prior treatment with an ERK1/2 inhibitor.
4. Prior major surgery within 28 days of the first dose of study treatment or minor surgical procedures ≤7 days.
5. Patients receiving unstable or increasing doses of corticosteroids.
6. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases.
7. Active infection including hepatitis B, and/or hepatitis C.
8. Known history of human immunodeficiency virus (HIV) infection.
9. Inadequate bone marrow reserve or organ function

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
AEs/SAEs | 18 months
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.

SECONDARY OUTCOMES:
Plasma concentrations | 18 months
  Venous blood samples for determination of total concentrations of ATG 017 in plasma to characterise the PK profile of ATG-017 for a particular dose level
Overall Response Rate (ORR) | 18 months
  To determine the overall response rate according to RECIST1.1, Chenson 2014, IWG 2003 and 2006
DOR | 18 months
  Duration of time from first occurrence of CR or PR until the first date that disease progression is objectively documented
Progression-Free Survival (PFS) | 18 months
  The time from the first dose date until disease progression or death from any cause

OTHER OUTCOMES:
Level of phospho-p90RSK | 18 months
  Blood samples will be analysed for the level of phospho-p90RSK
Level of transcript biomarker | 18 months
  Blood samples will be analysed for the level of DUSP6
Level of phospho-ERK | 18 months
  Blood samples will be analysed for the level of phospho-ERK
Level of total ERK | 18 months
  Blood samples will be analysed for the level of total ERK

CONTACTS AND LOCATIONS:
Overall Officials: Sai Lou, MD, Study Director — Clinical Research Physician; Anupa Kudva, MD, Study Director — Clinical Research Physician; Yiqiang Zhao, MD, Study Director — Executive Director
Locations (5):
- Australia (5):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Scientia Clinical Research, Randwick
  - Chris O'Brien Lifehouse, Sydney

IPD SHARING:
Plan to Share IPD: No